CLINICAL TRIAL: NCT00225693
Title: ELUTES III - V-Flex Plus PTX Drug Eluting Coronary Stent
Brief Title: V-Flex Plus PTX Drug Eluting Coronary Stent
Acronym: ELUTES III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 578
Record Dates: First submitted 2005-09-12; First posted 2005-09-26 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery; restenosis; patency; drug eluting; stent
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Device: drug eluting coronary stent

SUMMARY:
The study is intended to collect data to evaluate effectiveness and safety of drug eluting stent devices in a dose ranging assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be eligible to undergo planned treatment of a single de novo lesion in a native coronary artery.
* Patient must be an acceptable candidate for coronary artery bypass surgery
* Patient or legal guardian must have given informed consent
* Patient agrees to return at one month for an office visit to assess cardiovascular status and at 6 months for an office visit to assess cardiovascular status, an IVUS examination and a diagnostic angiogram.

Exclusion Criteria:

* Patient must be less than 18 years old
* Patient has history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* Patient is simultaneously participating in another investigative interventional cardiovascular device or drug study.
* Patient has known hypersensitivity or contraindication to aspirin, clopidogrel, or stainless steel, or a sensitivity to contrast dye.
* Women of child bearing potential.
* Patient has other medical condition that any cause non-compliance with the protocol, confound the results or is associated with limited life expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-10; Study Completion 2005-07

PRIMARY OUTCOMES:
Evaluation by IVUS of % diameter stenosis at follow up.

SECONDARY OUTCOMES:
Major adverse events
Target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Dens, MD, Principal Investigator — UZ Gasthuisberg Leuven
Locations (1):
- Contact Sponsor, Bloomington, Indiana, United States